CLINICAL TRIAL: NCT01311856
Title: Telephone Counseling-Mailed Materials Versus Internet Weight Management Interventions in Overweight Cancer Survivors
Brief Title: Telephone Counseling-Mailed Materials Versus Internet Interventions in Overweight Cancer Survivors
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-0504
Record Dates: First submitted 2011-03-04; First posted 2011-03-10 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer; Colorectal Cancer; Prostate Cancer
Keywords: Behavioral intervention; Exercise; Physical Assessment; Questionnaire; Survey; Telephone counseling; Internet interventions; Overweight cancer survivors; Exercise and weight management program
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms; Motor Activity | interventions — Surveys and Questionnaires; Exercise; Diet

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard Arm (mail/telephone)
  Interventions: Behavioral: Standard Arm (mail/telephone); Behavioral: Surveys and Questionnaires; Behavioral: Exercise and Diet
- Internet Arm
  Interventions: Behavioral: Internet Arm; Behavioral: Surveys and Questionnaires; Behavioral: Exercise and Diet

INTERVENTIONS:
Behavioral: Standard Arm (mail/telephone) — Participants will receive print materials on diet and exercise, telephone counseling calls (3 weekly calls, 2 semi-weekly calls, 4 monthly calls; 15-30 minutes in length), and customized mailed progress reports every 6 weeks to adhere to diet and exercise recommendations.
  Groups: Standard Arm (mail/telephone)
Behavioral: Internet Arm — Participants will access print information online. Participants will also participate in a discussion forum facilitated by the intervention staff, have the opportunity to email questions directly to the intervention staff, and receive progress reports every 6 weeks by email.
  Groups: Internet Arm
Behavioral: Surveys and Questionnaires — 9 online surveys to be completed before intervention sessions. After 14 weeks on study, questionnaires will be mailed for completion at home and mailed back to the study staff.
Behavioral: Exercise and Diet — 15 minutes of strength exercise every other day, >30 minutes of walking or other moderate-intensity exercise on 5 or more days of the week. Diet recommendations for both groups.

SUMMARY:
The goal of this behavioral research study is to learn if an internet or phone based exercise and weight management program can help cancer survivors to lose weight and change their eating and exercise behavior.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will be asked questions about your physical activity to make sure you are eligible. If you are found to have any pre-existing medical or dietary conditions that may prevent you from participating in this study, you will be asked to have your physician complete a form about your health conditions. You will only be allowed to participate in this study if he or she feels it is safe for you to engage in moderate physical activity. After physician clearance, if applicable, you will be scheduled for study visits at the Behavioral Research and Treatment Center (BRTC) at MD Anderson where you will complete tasks to measure your physical functioning ability. Information about your cancer and treatment history will be collected from your medical records as part of this study.

First Study Visit:

During the week before your first visit to the BRTC, you will complete the following tasks at home:

* You will wear an accelerometer and record your physical activities and exercise in a daily diary. An accelerometer is a small device that you wear on your waist during the day. It records how active you are. The accelerometer and diary will be mailed to you ahead of time, and a study staff member will call you to remind you when to start wearing the accelerometer and recording information in the daily diary.
* You will complete questionnaires that ask about any usual physical activities you may participate in, your health history, your quality of life, your social support, and your confidence for changing your eating and exercise behavior. The questionnaires will be mailed to you with the accelerometer and diary. You will complete the questionnaires at home when you have time. These questionnaires should take you no longer than about 30 minutes total to complete.
* Within a week of your first visit to the BRTC, you will complete 2 online "24-hour diet recalls", 1 during a weekday and the other on a weekend day. One of the diet recalls will be done during your first visit to the BRTC and the other will be done at your home. This involves completing an online questionnaire that asks about what you eat and drink. You will report everything you have consumed in the last 24 hours (from midnight to midnight). A study staff member will call you and tell you when to complete each 24-hour diet recall. Each phone call should last no longer than about 5 minutes, depending on if you have any questions for the study staff member.

You will bring the accelerometer, daily diary, and completed questionnaires with you to your first visit to the BRTC.

During your first visit to the BRTC, the following tests and procedures will be performed:

* You will complete any of the questionnaires that you may not have had time to complete at home.
* Your blood pressure, height, weight, and waist and hip measurements will be recorded.

You will also complete 5 simple performance tests that are designed to measure your aerobic function, lower body strength, upper body strength, agility (ability to move quickly), balance, and endurance:

* To test your aerobic fitness, you will complete a 2 minute step test. You will step in place. You must lift your leg up to midway between the knee and hip bone with each step. Your goal is to complete as many steps as possible within 2 minutes.
* To test your lower body strength, you will complete a 30 second chair-stand test. You will rise to an upright standing position from a fully seated position and then return to a fully seated position. You will repeat this as many times as you can within 30 seconds.
* To test your upper body strength, you will complete a timed arm-curl test. You will hold a dumbbell in each hand and slowly curl your arm up towards your shoulder, then slowly lower it until your arm is extended. You will repeat this with your other arm. You will complete this as many as you can within 30 seconds.
* To test your agility and balance, you will complete the "8 foot up-and-go test." For this test, you will sit in a chair facing a cone that marks exactly 8 feet from the chair. You will start the test sitting in the chair. When instructed to start, you will stand up and walk as fast as you can around the cone (without running or hitting the cone) and return to a fully seated position in the chair. You will repeat this test 2 times.
* Finally, you will complete a 6-minute walk test to measure your endurance. To complete this test, you will walk as fast as you can in an indoor hallway for 6 minutes. The distance you walk will be recorded.

A study staff member will instruct you on how to complete each of these tests correctly and safely. You will be given a chance to practice each test, except for the 6 minute walk test. If you have any physical problem or condition that you think may interfere with completing any of the tests, you should tell the study staff member right away.

Additionally, you will complete a dual energy x-ray absorptiometry (DEXA) scan to evaluate body composition. The DEXA scan exposes your body to radiation. The radiation you will receive is about a 10th of the radiation of a chest x-ray. If you are female, you will be asked if you are pregnant. If you state that you are not pregnant, you will receive the DEXA. If you are not sure if you are pregnant, you will have a urine pregnancy test done. If you are pregnant, you will not be able to take part in this study.

The visit to the BRTC should take approximately 2 1/2 hours to complete.

Internet and Phone Intervention Groups:

After you have completed your first visit to the BRTC, you will be randomly assigned (as in a toss of the dice) to either the internet-based intervention group or the phone-based intervention group. Each intervention program will take 6 months to complete. Two (2) out of 3 participants will be assigned to the internet group, and 1 out of 3 participants will be assigned to the phone group.

If you are assigned to the Internet Group:

* You will be given instructions on how to access the diet and exercise information online (www.WalkingSpree.com) that will help you to monitor the amount of fat grams and calories you eat.
* You will participate in a discussion group online that will be led by the study staff.
* You will be able to email questions directly to the study staff at any time.
* You will also receive personalized reports about your progress in meeting the diet and exercise recommendations every 6 weeks by email from the study staff. This is to help you to stay on track with the exercise and diet recommendations.

If you are assigned to the Phone Group:

* You will be given a fat gram and calorie counter to help you to monitor your eating habits.
* You will be given a binder of printed materials with information to help increase your exercise behavior and eat a more healthy diet.
* You will receive 1 counseling phone call each week for the first 3 weeks, then 1 call every 2 weeks for one month, and then 1 call each month for 4 months after that. Each phone call should last about 15-30 minutes. The calls will be recorded and reviewed by the research staff to make sure that the meetings are covering the program content.
* You will also receive personalized reports about your progress in meeting the diet and exercise recommendations every 6 weeks by mail from the study staff. This is to help you to stay on track with the exercise and diet recommendations.

Both groups will receive the following:

* You will receive a pedometer, which is a small device you wear on your belt that counts the number of steps you take. You will need to wear the pedometer all day (from when you wake up to when you go to sleep). You will need to record your daily steps either online or in the binder, depending on which group you are in.
* You will receive resistance bands, which are long, flexible, rubber bands with handles on each end that are used for resistance training. You will be given instructions with pictures, either online or in the binder, that tell and show you how to use the resistance bands correctly and safely. If you have any questions about using the resistance bands, you should email the study staff or call the study counselor, depending on which group you are assigned to.
* You will receive a portion guidance plate, which you are asked to use while eating to help you learn correct portion sizes.
* You will be provided with recommended goals for your exercise, diet, and weight.

After you have been on study for 14 weeks, questionnaires will be mailed to you to complete at home and mail back to the study staff. The questionnaires will ask about your level of physical activity, quality of life, and personal beliefs related to exercising and eating a healthy diet. The questionnaire should take about 20 minutes to complete.

You will also complete 9 online surveys before your intervention sessions while you are on study. These surveys will ask for information about your exercise and eating habits, as well as your personal beliefs related to changing exercise and dieting behavior. This information will help the study staff to give program related information that is specifically designed for you. The surveys should take about 5 minutes to complete.

Second Study Visit:

You will have a second study visit 6 months after the first visit. During the week before your second visit to the BRTC:

* You will wear an accelerometer for a week, record your physical activities and exercise in a daily diary, and complete the same questionnaires. The accelerometer, daily diary, and questionnaires will be mailed to you ahead of time.
* You will also complete 2 more online "24-hour diet recalls" within a week of your second visit. A study staff member will call you and tell you when to complete each diet recall.

You will bring the accelerometer, daily diary, and completed questionnaires with you to your second visit to the BRTC.

During your second visit to the BRTC:

* You will complete any of the questionnaires that you may not have had time to complete at home.
* Your blood pressure, weight, and waist and hip measurements will be recorded.
* You will complete the 5 simple performance tests and a DEXA scan (after testing negative for pregnancy, if applicable).

Length of Study:

You will remain on study for up to 6 months after your first visit to the BRTC.

This is an investigational study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of either loco-regional breast cancer (Stages 0 - IIIA), colon cancer (Stages I - II), endometrial cancer (Stages I - IIIa) or prostate cancer (Stages I - II);
2. No history of other cancers (excluding non-melanoma skin cancer);
3. Age 18 years of age or older;
4. BMI greater than or equal to 25;
5. Has access to a computer with high-speed internet;
6. Has access to a telephone for possible multiple counseling sessions;
7. Living in the Houston area (Harris county or a contiguous county);
8. Has agreed in the protocol 2009-0544 survey to be re-contacted about studies (for breast, prostate, and colon cancer survivors), or is an endometrial cancer survivor seen seen by an MD Anderson gynecologic oncologist at MD Anderson or an outreach site;
9. Able to come to MD Anderson for assessments at baseline and six-month intervals;
10. Has completed primary cancer treatment and is at least 3 months from surgery (if elected);
11. Able to read and speak English; and
12. Able to provide informed consent.

Exclusion Criteria:

1. Have pre-existing medical conditions that preclude adherence to an unsupervised exercise program or a low-fat, high fruit and vegetable (F&V) diet;
2. Persons using walker or wheelchair/scooter;
3. Women who are pregnant; and
4. Patients that are identified as having metastatic disease at the time of recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants recruited from UT MD Anderson Cancer Center clinics in Houston, Texas
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-03 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | 6 months
  Recruitment and drop-out rates in both treatment groups used to assess internal validity of study by comparison of drop-out between two study conditions, and drop-outs to completers.

SECONDARY OUTCOMES:
Drop-Out Rate | 6 months
  Recruitment and drop-out rates in both treatment groups used to assess internal validity of study by comparison of drop-out between two study conditions, and drop-outs to completers.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Basen-Engquist, PHD, BA, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Cox M, Basen-Engquist K, Carmack CL, Blalock J, Li Y, Murray J, Pisters L, Rodriguez-Bigas M, Song J, Cox-Martin E, Demark-Wahnefried W. Comparison of Internet and Telephone Interventions for Weight Loss Among Cancer Survivors: Randomized Controlled Trial and Feasibility Study. JMIR Cancer. 2017 Sep 27;3(2):e16. doi: 10.2196/cancer.7166. PMID 28954716
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org